CLINICAL TRIAL: NCT05444751
Title: Evaluating General Anesthesia With Erector Spinae Plane Block vs. Spinal Anesthesia With Erector Spinae Plane Block in Lumbar Decompression Surgeries
Brief Title: GA + ESP vs. SA + ESP in Lumbar Decompression Surgeries
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-2478
Record Dates: First submitted 2022-06-20; First posted 2022-07-06 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-01

CONDITIONS: Lumbar Disc Herniation; Lumbar Disc Disease; Lumbar Radiculopathy
Keywords: Degenerative Disc Disease; Lumbar Spine
MeSH Terms: conditions — Intervertebral Disc Displacement; Intervertebral disc disease; Radiculopathy; Intervertebral Disc Degeneration | interventions — Anesthetics, General; Parapsychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SA + ESP Block (Experimental): Spinal Anesthesia: Patients will be provided with iv sedation, if desired, to facilitate placement of spinal anesthetic. Midazolam (2-5mg, iv), ketamine (up to 20 mg, lv) and/or propofol (0.1-0.2 mg/kg) will be permitted.
  Interventions: Drug: SA + ESP
- GA + ESP Block (Active Comparator): General anesthesia: induction of general anesthesia to facilitate endotracheal intubation: fentanyl (up to 2μg.kg.min-1), propofol (1-2 mg.kg-1), vecuronium (1-2 mg.kg-1).
  Interventions: Drug: General anesthetic

INTERVENTIONS:
Drug: General anesthetic — Maintenance of general anesthesia: propofol infusion (50-150 μg.kg.min-1); ketamine infusion (up to 50 mg total); and inhaled anesthetic agent (isoflurane or sevoflurane) up to 0.5 MAC. N20 is not permitted.
  Emergence from general anesthesia: N20 may be used during closure of the surgical incision to facilitate rapid emergence.
  Other Names: GA + ESP
  Arms: GA + ESP Block
Drug: SA + ESP — The choice of local anesthetic for spinal anesthesia will be confirmed after consultation with the attending surgeon to determine duration of surgery. For expected surgical times less than 90 minutes, up to 4 mL 1.5% mepivacaine (60 mg) will be used. Where the anticipated surgical duration is longer than 90 minutes, 2 mL 0.5% bupivacaine (10 mg) may be substituted. After patient (prone) positioning, maintenance of sedation will be achieved with a target RASS score of 0 to -1.
  Propofol (25-50 μg.kg.min-1) and ketamine (up to 50 mg total dose) infusions will be titrated to effect. Intermittent boluses of propofol (10-20mg) may be used to achieve the desired sedation, as needed.
  Patients will be offered to option of awake surgery, where no sedation will be provided, if preferred. Patients will be informed that at any time before or during the procedure, they may change their mind, and receive sedation.
  Other Names: Erector Spinae Block
  Arms: SA + ESP Block

SUMMARY:
The purpose of this study is to determine the optimal anesthetic routine for lumbar decompression surgery. General Anesthesia is the standard of care in spine surgery. Spinal anesthesia in decompressive procedures can be the new standard of care. Recently, it has been found that regional analgesia is option that has been shown to improve pain and opioid-related outcomes after spine surgery, but has not yet been studied in combination with spinal anesthesia. This is study that consists of two groups: standard of care general anesthesia with a nerve block and a spinal anesthesia with nerve block. Patients are randomized to either of the two groups. There will be 71 patients enrolled in each group for this study.

DETAILED DESCRIPTION:
An early comparative analysis between GA and SA in spine surgery explored perioperative effects of the technique on cost and satisfaction among patients, anesthesiologists, and surgeons. Patients who underwent surgery under SA had better outcomes, including hemodynamic stability, shorter hospitalization time, and shorter time to return to work. Postoperatively, SA was associated with lower numeric pain rating scale (NPRS) scores and earlier time to mobilization and first oral intake. Moreover, SA had lower costs and higher reported satisfaction among patients, surgeons, and anesthesiologists.

Subsequent studies have consistently concluded that SA is associated with shorter surgical duration and less blood loss in patients compared to GA for spine surgery. Additionally, hospital length of stay has been reported to be shorter after SA, perhaps due to lower incidence of complications found in several series.

Early postoperative pain control may also be superior after SA in patients undergoing microdiscectomy, attributed to residual sensory block after SA. In addition to higher peaks in pain scores and significantly greater analgesic requirements among the GA group, more episodes of nausea were described, and more antiemetic medications were given.

Intraoperative neurophysiological monitoring (IONM) during procedures such as one and two-level microdiscectomies and laminotomies, use somatosensory evoked potentials (SSEPs), motor evoked potentials (MEPs), and electromyograms (EMGs) as routine during surgery. Surgeons can monitor spinal cord and nerve root function in real-time, take measures to prevent/lessen irritation or potential damage and can detect intraoperative neurologic injuries. Microdiscectomies and laminotomies are one of the most common spinal procedures, which can be performed in both its "open" and "minimally invasive" variations, is a well-established, safe procedure. However, studies have shown that the use of IONM in smaller, less complicated procedures such as microdiscectomies or laminotomies, may add to the overall cost without providing many benefits. Decompressive surgeries under SA cover only the spine and nerve roots within a specific region. Subsequently, SA does not transmit sensory impulses to the brain, therefore, neuromonitoring such as somatosensory evoked potentials (SSEPs) are not required in cases such as these. Certain types of IOMN can be performed under GA, as transmissions of sensory impulses are sent to the brain to identify neural irritation or injury and define the nature of the injury, which will allow the surgeon to complete the procedure without risking further injury.

Despite broad patient acceptance of SA for lower extremity procedures, and abundant evidence to support superior outcomes after orthopedic surgery, SA has never gained wide acceptance in lumbar spine surgery. Arguments against SA for lumbar decompression surgeries include the potential for airway complications in sedated prone positioned patients, the possibility for neural injury if an awake patient moves during decompressive procedures, the potential for intraoperative conversion to GA due to insufficient duration or failed SA, and confounding of the early postoperative neurologic examination.

The Erector Spinae Plane Block (ESP) is a novel fascial plane block, originally described as an effective treatment for thoracic neuritis. Since its first description, the ESP block has been applied to a broad range of surgical procedures, with benefits for opioid-sparing analgesia, a good safety profile, and few complications. The ESP block is considered to be relatively easy to perform when compared to other thoracic or neuraxial blocks, such as epidural and paravertebral blocks. The clinical findings of early studies have been supported by anatomical studies in cadavers demonstrating the appropriate spread of local anesthetic to the dorsal and ventral rami of the nerve roots of the thoracic spine.

The value of ESP block for spine surgery has likewise been suggested in case reports case series, and retrospective cohort studies. Each concludes significant opioid-sparing capacity and improved NRS pain scores in patients who receive ESP blocks for a variety of spine surgery procedures.

More recently, results from 2 RCTs describing outcomes after ESP block for lumbar decompression have been reported. In the first, 60 patients were randomized to receive bilateral ESPB or no intervention. NRS scores and tramadol consumption were significantly lower in the first 24 hours after surgery, and the time to requesting opioid analgesia was significantly longer in patients were received ESPB. In the second RCT, postoperative morphine consumption was lower in patients who received ESPB compared to patients who did not receive ESPB. NRS scores were lower up to 6 hours after surgery in the ESPB group, and patient satisfaction scores were higher

HSS anesthesiologists have been offering ESP blocks for spine surgery via posterior approach since 2017. A recent retrospective analysis of over 800 patients at HSS supports ESP blocks as analgesic and opioid-sparing in our spine surgery population.

As the above literature review suggests, there is unmet clinical and research need to explore the optimal anesthetic-analgesic regimen in patients undergoing minimally invasive lumbar decompression. This study has the potential to address the risk, benefits advantages and disadvantages of SOC GA for patients undergoing spine surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the ages 18- 80 years
* Patients with one or two-level microdiscectomy, laminotomy, or foraminotomy - prior spine surgery is allowed only if surgery was preformed at other levels.
* Able to follow study protocol
* Able to provide informed consent

Exclusion Criteria:

* Surgery with planned need for postoperative surgical drain.
* Allergies of contraindication to any study anesthetic or analgesic medications.
* Morbid obesity, defined as BMI > 35 kg/m2.
* Involved in the study of another investigational product that may affect the outcome.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
QoR15 survey scores | The QoR15 survey will be assessed preoperatively (in holding area). It will be assessed again immediately after surgery in the PACU and then at 2-weeks postoperatively at the patient's first follow-up visits
  The primary outcome is the difference in the quality of recovery-15 (QoR15) score between the groups at each timepoint (before surgery, after surgery, and at their first 2 week follow-up visit). For this survey, a high number represents something that occurs often, while a low number indicates something that rarely or never occurs. Depending on the category/question asked, this may be good or bad. The questions on the survey will be split and compared so that for one subset of questions a high number is good while the opposite is true for the other subset of questions. This will be done so the comparison between groups is more accurate and meaningful.

SECONDARY OUTCOMES:
NRS Survey Pain Scores | The NRS will be assessed preoperatively (in holding area), postoperatively in PACU, and 2 weeks postoperatively at the patient's first follow-up
  Numeric rating scale (NRS) survey will be asked in holding (before surgery), in the PACU (after surgery), and at the patients first 2week follow-up visit. Most patients will be discharged a few hours after waking up, barring no complications, therefore may only be assessed the NRS survey immediately after surgery (same as QoR15). For this scale (0-10), a higher number indicates more pain in that specified body part, while a lower score indicates little or no pain in that body part.
Opioid Consumption | From surgery through 24 hours postoperatively
  Opioid consumption will be tracked intraoperatively and total from PACU arrival to 24 hours surgery
Anesthetic(s) Time | Intraoperatively
  induction (from induction to anesthesia-ready), emergence (from surgery-end to out-of-OR for SA group; and from surgery-end to extubation for GA groups); duration of SA (from placement to resolution).
Surgical Duration | Intraoperatively
  Time of surgery will be compared between groups from skin incision to skin closure
Complications | Length of stay at the hospital (up to 3 days postoperatively)
  nausea, vomiting, urinary retention, escalation to a higher level of postoperative care, conversion from SA to GA, neurologic (extremity numbness, weakness, paresthesia).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLain RF, Kalfas I, Bell GR, Tetzlaff JE, Yoon HJ, Rana M. Comparison of spinal and general anesthesia in lumbar laminectomy surgery: a case-controlled analysis of 400 patients. J Neurosurg Spine. 2005 Jan;2(1):17-22. doi: 10.3171/spi.2005.2.1.0017. PMID 15658121
- [Background] Kilic ET, Naderi S. Effects of Anesthesia Protocol on Perioperative Outcomes and Costs of Lumbar Microdiscectomies. Turk Neurosurg. 2019;29(6):843-850. doi: 10.5137/1019-5149.JTN.25737-18.4. PMID 30984998
- [Background] Melvin JP, Schrot RJ, Chu GM, Chin KJ. Low thoracic erector spinae plane block for perioperative analgesia in lumbosacral spine surgery: a case series. Can J Anaesth. 2018 Sep;65(9):1057-1065. doi: 10.1007/s12630-018-1145-8. Epub 2018 Apr 27. PMID 29704223
- [Background] Marks R. Keeping patient awake during spine surgery is cutting recovery time in half. https://www.ucsf.edu/news/2019/03/413446/spine-surgery-while-patients-are-awake-speeds-healing Accessed 1/24/2020
- [Background] Harbers C. Duke spine surgeon offers awake surgery to patients. https://medschool.duke.edu/about-us/news-and-communications/som-magnify/duke-spine-surgeon-offers-awake-surgery-patients Accessed 1/24/2020
- [Background] Kara I, Celik JB, Bahar OC. Comparison of spinal and general anesthesia in lumbar disc surgery. Journal of Neurological Sciences (Turkish) 28:487-496, 2011 9.
- [Background] McLain RF, Tetzlaff JE, Bell GR, Uwe-Lewandrowski K, Yoon HJ, Rana M. Microdiscectomy: spinal anesthesia offers optimal results in general patient population. J Surg Orthop Adv. 2007 Spring;16(1):5-11. PMID 17371640
- [Background] Meng T, Zhong Z, Meng L. Impact of spinal anaesthesia vs. general anaesthesia on peri-operative outcome in lumbar spine surgery: a systematic review and meta-analysis of randomised, controlled trials. Anaesthesia. 2017 Mar;72(3):391-401. doi: 10.1111/anae.13702. Epub 2016 Oct 22. PMID 27770448
- [Background] Dagistan Y, Okmen K, Dagistan E, Guler A, Ozkan N. Lumbar Microdiscectomy Under Spinal and General Anesthesia: A Comparative Study. Turk Neurosurg. 2015;25(5):685-9. doi: 10.5137/1019-5149.JTN.10300-14.1. PMID 26442531
- [Background] Demirel CB, Kalayci M, Ozkocak I, Altunkaya H, Ozer Y, Acikgoz B. A prospective randomized study comparing perioperative outcome variables after epidural or general anesthesia for lumbar disc surgery. J Neurosurg Anesthesiol. 2003 Jul;15(3):185-92. doi: 10.1097/00008506-200307000-00005. PMID 12826965
- [Background] Dhall S, Gonzalez A, Jallo G, et al.
- [Background] Krause KL, Cheaney Ii B, Obayashi JT, Kawamoto A, Than KD. Intraoperative neuromonitoring for one-level lumbar discectomies is low yield and cost-ineffective. J Clin Neurosci. 2020 Jan;71:97-100. doi: 10.1016/j.jocn.2019.08.116. Epub 2019 Sep 5. PMID 31495654
- [Background] Pajewski TN, Arlet V, Phillips LH. Current approach on spinal cord monitoring: the point of view of the neurologist, the anesthesiologist and the spine surgeon. Eur Spine J. 2007 Nov;16 Suppl 2(Suppl 2):S115-29. doi: 10.1007/s00586-007-0419-6. Epub 2007 Jul 10. PMID 17619913
- [Background] Memtsoudis SG, Cozowicz C, Bekeris J, Bekere D, Liu J, Soffin EM, Mariano ER, Johnson RL, Hargett MJ, Lee BH, Wendel P, Brouillette M, Go G, Kim SJ, Baaklini L, Wetmore D, Hong G, Goto R, Jivanelli B, Argyra E, Barrington MJ, Borgeat A, De Andres J, Elkassabany NM, Gautier PE, Gerner P, Gonzalez Della Valle A, Goytizolo E, Kessler P, Kopp SL, Lavand'Homme P, MacLean CH, Mantilla CB, MacIsaac D, McLawhorn A, Neal JM, Parks M, Parvizi J, Pichler L, Poeran J, Poultsides LA, Sites BD, Stundner O, Sun EC, Viscusi ER, Votta-Velis EG, Wu CL, Ya Deau JT, Sharrock NE. Anaesthetic care of patients undergoing primary hip and knee arthroplasty: consensus recommendations from the International Consensus on Anaesthesia-Related Outcomes after Surgery group (ICAROS) based on a systematic review and meta-analysis. Br J Anaesth. 2019 Sep;123(3):269-287. doi: 10.1016/j.bja.2019.05.042. Epub 2019 Jul 24. PMID 31351590
- [Background] Attari MA, Mirhosseini SA, Honarmand A, Safavi MR. Spinal anesthesia versus general anesthesia for elective lumbar spine surgery: A randomized clinical trial. J Res Med Sci. 2011 Apr;16(4):524-9. PMID 22091269
- [Background] Greenbarg PE, Brown MD, Pallares VS, Tompkins JS, Mann NH. Epidural anesthesia for lumbar spine surgery. J Spinal Disord. 1988;1(2):139-43. PMID 2980070
- [Background] Hassi N, Badaoui R, Cagny-Bellet A, Sifeddine S, Ossart M. [Spinal anesthesia for disk herniation and lumbar laminectomy. Apropos of 77 cases]. Cah Anesthesiol. 1995;43(1):21-5. French. PMID 7671051
- [Background] Jellish WS, Thalji Z, Stevenson K, Shea J. A prospective randomized study comparing short- and intermediate-term perioperative outcome variables after spinal or general anesthesia for lumbar disk and laminectomy surgery. Anesth Analg. 1996 Sep;83(3):559-64. doi: 10.1097/00000539-199609000-00021. PMID 8780281
- [Background] Riegel B, Alibert F, Becq MC, Duckert I, Krivosic-Horber R. [Lumbar disk herniation with surgical option: general versus local anesthesia. Round table]. Agressologie. 1994;34 Spec No 1:33-7. French. PMID 7818012
- [Background] Tetzlaff JE, Baird BA, Yoon HJ. Spinal anesthesia with plain bupivicaine for lumbar spine surgery. Can J Anaesth. 1990 May;37(4 Pt 2):S61. No abstract available. PMID 2361303
- [Background] Tetzlaff JE, O'Hara J, Bell G, Grimm K, Yoon HJ. Influence of baricity on the outcome of spinal anesthesia with bupivacaine for lumbar spine surgery. Reg Anesth. 1995 Nov-Dec;20(6):533-7. PMID 8608073
- [Background] Koekemoer AM, Henkel C, Greenhill LJ, Dey A, van Breugel W, Codella C, Antonucci R. A water-vapour giga-maser in the active galaxy TXFS2226-184. Nature. 1995 Dec 14;378(6558):697-9. doi: 10.1038/378697a0. PMID 7501016
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Brandão J, Mamôru T: Sakae Erector Spine Plane Block in Different Surgeries. J Anes Perio Manag 4: 005
- [Background] Almeida CR, Oliveira AR, Cunha P. Continuous Bilateral Erector of Spine Plane Block at T8 for Extensive Lumbar Spine Fusion Surgery: Case Report. Pain Pract. 2019 Jun;19(5):536-540. doi: 10.1111/papr.12774. Epub 2019 Mar 15. PMID 30758122
- [Background] Chin KJ, Lewis S. Opioid-free Analgesia for Posterior Spinal Fusion Surgery Using Erector Spinae Plane (ESP) Blocks in a Multimodal Anesthetic Regimen. Spine (Phila Pa 1976). 2019 Mar 15;44(6):E379-E383. doi: 10.1097/BRS.0000000000002855. PMID 30180150
- [Background] Singh S, Chaudhary NK. Bilateral Ultasound Guided Erector Spinae Plane Block for Postoperative Pain Management in Lumbar Spine Surgery: A Case Series. J Neurosurg Anesthesiol. 2019 Jul;31(3):354. doi: 10.1097/ANA.0000000000000518. No abstract available. PMID 29965831
- [Background] Ueshima H, Inagaki M, Toyone T, Otake H. Efficacy of the Erector Spinae Plane Block for Lumbar Spinal Surgery: A Retrospective Study. Asian Spine J. 2019 Apr;13(2):254-257. doi: 10.31616/asj.2018.0114. Epub 2018 Nov 15. PMID 30424594
- [Background] Yayik AM, Cesur S, Ozturk F, Ahiskalioglu A, Ay AN, Celik EC, Karaavci NC. Postoperative Analgesic Efficacy of the Ultrasound-Guided Erector Spinae Plane Block in Patients Undergoing Lumbar Spinal Decompression Surgery: A Randomized Controlled Study. World Neurosurg. 2019 Jun;126:e779-e785. doi: 10.1016/j.wneu.2019.02.149. Epub 2019 Mar 8. PMID 30853517
- [Background] Singh S, Choudhary NK, Lalin D, Verma VK. Bilateral Ultrasound-guided Erector Spinae Plane Block for Postoperative Analgesia in Lumbar Spine Surgery: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Oct;32(4):330-334. doi: 10.1097/ANA.0000000000000603. PMID 31033625
- [Background] Soffin et al, 2021, in prep, personal communication